CLINICAL TRIAL: NCT04419142
Title: Total Infrapatellar Fat Pad Excision Leads to Worse Isokinetic Performance in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Total Fat Pad Excision Leads to Worse Isokinetic Performance in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Erdem A Sezgin, Co-Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1464/2017
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee; Knee Arthritis
Keywords: Infrapatellar fat pad; Total knee arthroplasty; Isokinetic test; Strength
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients were randomized in a 1:1 ratio via computer-generated randomization using Microsoft Excel 2016 (Microsoft Corporation, Seattle, WA, USA) to be allocated in the total or partial infrapatellar fat pad excision group before the TKA operation (Figure 1). Unblinded senior resident implemented the randomization. Patients and physiatrists performing isokinetic measurements were blinded to group allocation.
Who Masked: Participant, Investigator
Masking Description: Patients and physiatrists performing isokinetic measurements were blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total infrapatellar fat pad excision group (Experimental): Infrapatellar fat pad was totally excised during total knee arthroplasty in patients randomized to this group.
  Interventions: Procedure: Total infrapatellar fat pad excision
- Partial infrapatellar fat pad excision group (Experimental): Infrapatellar fat pad was partially excised during total knee arthroplasty in patients randomized to this group.
  Interventions: Procedure: Partial infrapatellar fat pad excision

INTERVENTIONS:
Procedure: Total infrapatellar fat pad excision — Exposure for total knee arthroplasty (TKA) commonly includes total excision of the infrapatellar fat pad (IPFP). The rationale behind this is to obtain improved access to the lateral tibial plateau allowing a more accurate bone cut, baseplate placement and easier management of soft tissue interposition in the bone and cement interface. However, there is growing concern that as the IPFP is a highly vascularized and innervated fibrous adipose tissue filling the anterior compartment of the knee, its complete excision may have a detrimental effect on knee biomechanics and ultimately, TKA outcome. The reason for this effect has been suggested to be patellar tendon (PT) scarring and shortening via ischemic contracture following impaired vascularization, maintenance and biological repair of the tendon.
  Arms: Total infrapatellar fat pad excision group
Procedure: Partial infrapatellar fat pad excision — It has been suggested in the literature that partial infrapatellar fat pad excision instead of total excision would diminish the potential negative effect on patellar tendon and knee biomechanics. However, there is only limited data in the literature and choice of total/partial infrapatellar fat pad excision in TKA remains debatable.
  Arms: Partial infrapatellar fat pad excision group

SUMMARY:
There are concerns that total infrapatellar fat pad (IPFP) excision in total knee arthroplasty (TKA) results in patellar tendon shortening due to ischemic contracture. But, individual preference of the surgeon is still the main determinant between total or partial excision. The aim of this randomized controlled trial is to compare knee society score (KSS), knee extension and flexion peak torque in patients undergoing TKA with total IPFP excision or partial IPFP excision. The hypothesis of the study is that during TKA, total IPFP excision would lead to worse isokinetic performance and clinical outcome.

A total of 72 patients scheduled to undergo TKA for primary osteoarthritis of the knee by a single surgeon were randomly assigned to either the total or partial excision group. Patients were evaluated preoperatively and at postoperative 1 year, with Knee Society Score (KSS) and isokinetic measurements. Physiatrist doing isokinetic tests and patients were blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 80 years
* Scheduled to undergo unilateral TKA on for primary knee osteoarthritis

Exclusion Criteria:

* Inflammatory arthritis
* Post-traumatic osteoarthritis
* Previous knee surgery
* Neuromuscular diseases
* Bilateral TKA
* Insufficiency of collateral ligaments

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Peak knee extensor torque change from baseline to postoperative 12 months | Preoperative - Postoperative 12 months
  Change in peak knee extensor torque from baseline (preoperatively) to 12 months post implantation was evaluated for the operated knee under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).
Peak knee flexor torque change from baseline to postoperative 12 months | Preoperative - Postoperative 12 months
  Change in peak knee flexor torque from baseline (preoperatively) to 12 months post implantation was evaluated for the operated knee under the supervision of the same physiatrist. The Isokinetic measurements were performed using a Biodex System III Isokinetic Dynamometer, version 3.03 (Biodex Medical Inc.,Shirley, NY, USA). Concentric isokinetic knee flexion-extensions were assessed at a preset velocity of 60º/sec, over a range of motion of 0º to 110º for both parameters. A fixed number of 10 flexion-extension repetitions was completed by each patient. Torque was assessed in Newton-meters (N m).

SECONDARY OUTCOMES:
Knee Society Score (KSS) change from baseline to postoperative 12 months | Preoperative - Postoperative 12 months
  Change in the Knee Society Score from baseline (preoperatively) to 12 months post implantation was evaluated.
  The Knee Society Score (KSS) is comprised to two sections (each worth 100 points) for a maximum 200 points. One section is the Knee Society Clinical Score (KSCS) - points are given for pain, motion, and stability and points are deducted for flexion contracture, extension lag, and misalignment. The other section is the Knee Society Functional Score (KSFS) - points are assigned for walking distances and climbing stairs and points are deducted for use of walking aids. For each section, a score of 80-100 = excellent, 70-79 = good; 60-69 = fair; and < 60 = poor.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Çankaya, MD, Principal Investigator — Aksaray University Training and Research Hospital
Locations (1):
- Aksaray University Training and Research Hospital, Aksaray, Turkey (Türkiye)